CLINICAL TRIAL: NCT04815824
Title: Comparison of Exercise Mode on Disruptions in Calcium Homeostasis
Brief Title: Exercise Mode and Acute Bone Resorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: F3593-P; 1I21RX003593 (NIH)
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Osteoporosis; Aging
Keywords: exercise; bone resorption; calcium
MeSH Terms: conditions — Osteoporosis; Motor Activity; Bone Resorption

STUDY DESIGN:
Intervention Model Description: Crossover design comparing mode of endurance exercise (cycling versus treadmill).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stationary Cycling (Experimental): All participants will complete one, 60-minute bout of stationary cycling
  Interventions: Behavioral: Exercise Mode
- Treadmill Walking (Experimental): All participants will complete one, 60-minute bout of treadmill walking
  Interventions: Behavioral: Exercise Mode

INTERVENTIONS:
Behavioral: Exercise Mode — Stationary cycling or treadmill walking

SUMMARY:
Endurance exercise is often recommended to improve cardiometabolic health and maintain bone health throughout life and to prevent osteoporotic fracture. However, there is evidence to suggest that bone does not always adapt in the way that is expected, and that endurance exercise may lead to bone loss under certain conditions. Disruptions in calcium homeostasis during exercise may explain this observation, and preliminary data suggests that the mode of exercise (i.e., cycling versus treadmill) may result in different magnitudes of change in bone biomarkers. The purpose of this study is to determine if mode of exercise results in a differential bone biomarker response to an acute exercise bout in older Veterans. Blood samples will be collected before, during, and after 2 acute exercise bouts: 1) brisk treadmill walking; and 2) vigorous stationary cycling. Bouts will be matched for relative intensity and duration. This data will be used to develop future exercise interventions in older Veterans aimed at preserving both cardiometabolic and bone health.

DETAILED DESCRIPTION:
Endurance exercise is frequently recommended as a means to reduce the risk of cardiometabolic diseases and to reduce the risk of osteoporotic fracture. However, bone does not always adapt in the way that would be expected, and there is evidence that endurance exercise may lead to bone loss under certain conditions. It is the investigators contention that disruptions in calcium homeostasis during exercise, resulting in decreases in serum ionized calcium (iCa) and increases in parathyroid hormone (PTH) and c-telopeptide of type I collagen (CTX; a marker of bone resorption) at the onset of exercise, may be responsible for the lack of improvements in bone mineral density that are anticipated. Acute studies in this area have predominantly focused on young, healthy adults, primarily men, during stationary cycling exercise. Few studies have been conducted in older adults, but those studies have found that older adults experience similar disruptions in calcium homeostasis in response to an acute bout of endurance exercise. Preliminary comparisons of the investigators studies, as well as research from other labs, also suggests that that mode of exercise conducted during these acute exercise bouts may be an important determining factor in the catabolic bone response to exercise. It appears that weight-bearing exercise (i.e., treadmill) results in smaller increases in PTH and CTX compared to weight-supported exercise (i.e., stationary cycling). This has never been tested using a within-subjects design, so it is unclear if these observed differences are due to the mode of exercise, lab-to-lab differences, or other underlying factors. To address this gap in knowledge, 30 Veterans (15 men, 15 women), aged 60+ years, will complete two 1-hour acute exercise bouts: 1) brisk treadmill walking at 70-80% of maximal heart rate; 2) vigorous stationary cycling at 70-80% maximal heart rate. Blood samples will be collected to measure iCa, PTH, CTX and procollagen type I n-terminal propeptide (P1NP) before, during, and after each exercise bout. The order of the exercise bouts will be randomized and counter-balanced. The primary aim is to determine if mode of exercise results in a differential bone biomarker response in older Veterans. This information is essential for understanding how future exercise interventions should be designed to benefit both cardiometabolic health and bone health. This is especially relevant to Veteran health due to the high burden of both cardiometabolic diseases (e.g., diabetes, heart disease) in the population, as well as evidence of increased osteoporotic fracture risk. The proposed research is significant because it is addressing a knowledge gap that has prevented the ability to design exercise and lifestyle interventions aimed at preserving multiple components of Veteran health, which could have a lasting impact on Veteran quality of life and functional independence. The proposed research is innovative because it is testing a novel hypothesis, the mode of exercise on disruptions in calcium homeostasis, in a population that could greatly benefit from the knowledge to be gained. While the proposed research is an acute study, the results generated will be used to design future clinical interventions for Veteran health. Long-term, information gained from this research will help to define the optimal exercise prescription to improve cardiometabolic without compromising bone health aging Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy older (60+ y) Veteran women and men will be eligible to participate
* All volunteers must be accustomed to performing 60 minutes of vigorous cycling and treadmill exercise

Exclusion Criteria:

* impaired renal function, defined as an eGRF of <60 mL/min/1.73m2;(Florkowski and Chew-Harris 2011)
* hepatobiliary disease, defined as liver function tests (AST, ALT) >1.5 times the upper limit of normal
* thyroid dysfunction, defined as an ultrasensitive thyroid stimulating hormone (TSH) <0.5 or >5.0 mU/L
* serum Ca <8.5 or >10.3 mg/dL; 5) serum 25(OH)D <20 ng/mL
* uncontrolled hypertension, defined as resting systolic blood pressure (BP) >150 mmHg or diastolic BP >90 mmHg
* history of type 1 or type 2 diabetes
* cardiovascular disease; defined as subjective or objective indicators of ischemic heart disease (e.g., angina, ST segment depression) or serious arrhythmias at rest or during the graded exercise test (GXT)

  * volunteers who have a positive GXT can be re-considered after follow-up evaluation, which must include diagnostic testing (e.g., stress echocardiogram or thallium stress test) with interpretation by a cardiologist
* anemia, defined as a serum hemoglobin <12.1 g/dL for women and <14.3 g/dL for men
* fracture in the past 6 months
* current diagnosis or symptoms of COVID-19

  * In the event of abnormal BP, live function, TSH, 25(OH)D, or hemoglobin values, volunteers can be reassessed, including after appropriate follow-up evaluation and treatment by a primary care provider
  * Those who have experienced symptoms of COVID-19 or have been formally diagnosed will be allowed to participate once symptoms have resolved and they are approved to return to exercise by their primary care provider

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Wherry, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stationary Cycling First, Then Treadmill Walking: All participants will complete one, 60-minute bout of stationary cycling. Approximately one week later, participants will complete a 60-minute bout of treadmill walking.
- Treadmill Walking First, Then Stationary Cycling: All participants will complete one, 60-minute bout of treadmill walking. Approximately one week later, participants will complete a 60-minute bout of stationary cycling.
Period: First Intervention (60 Minutes)
Arm/Group | Stationary Cycling First, Then Treadmill Walking | Treadmill Walking First, Then Stationary Cycling
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Stationary Cycling First, Then Treadmill Walking | Treadmill Walking First, Then Stationary Cycling
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Second Intervention (60 Minutes)
Arm/Group | Stationary Cycling First, Then Treadmill Walking | Treadmill Walking First, Then Stationary Cycling
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Because all participants completed both interventions (60 minutes of stationary cycling, 60 minutes of treadmill walking), participant characteristics have been collapsed into one Arm/Group titled "All Study Participants."
Groups:
- All Study Participants: All participants complete both a stationary cycling and a treadmill walking exercise bout, but the order was randomized.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
Cardiorespiratory Fitness (VO2peak) [Mean (Standard Deviation); unit: mL/kg/min] | 25.8 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: C-telopeptide of Type I Collagen (CTX) Change
Description: CTX is a blood marker of bone resorption. Reference range is 0.1-0.8 ng/mL with lower concentrations suggesting less bone resorption.
Time Frame: Before to up to 48 hours after acute exercise bout
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Stationary Cycling | Treadmill Walking
Number analyzed (Participants) | 9 | 9
ng/mL | 0.09 (0.06) | 0.08 (0.07)

2. Secondary Outcome: Procollagen of Type I N-terminal Propeptide (P1NP) Change
Description: PINP is a blood marker of bone formation. Reference range is 19-80 ng/mL with lower concentrations suggesting less bone formation.
Time Frame: Before to up to 48 hours after acute exercise bout
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Stationary Cycling | Treadmill Walking
Number analyzed (Participants) | 9 | 9
ng/mL | -3.1 (7.8) | -1.5 (7.1)

ADVERSE EVENTS:
Time Frame: Adverse event information was collection from time of informed consent to completion of the study, which was approximately 8 weeks.
Arm/Group | Stationary Cycling | Treadmill Walking
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT04815824/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT04815824/ICF_000.pdf